CLINICAL TRIAL: NCT02051205
Title: Parkinson's Disease Registry（PDR）
Brief Title: Parkinson's Disease Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Shin-Yuan Chen, Department of Neurosurgery, Buddhist Tzu Chi General Hospital
Other Study IDs: TCRD-I102-03; TCRD-I102-03 (Other Grant/Funding Number: TCRD-I102-03)
Record Dates: First submitted 2013-10-30; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease, risk factors, epidemiology
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the Parkinson's disease Registry (PDR) is to develop a nation-wide database of persons with Parkinson's disease (PD) in Taiwan.

DETAILED DESCRIPTION:
Among degenerative neurological disease, PD is the second most common disorder. Although a wide range of incidence and prevalence rate exist in reviewed literatures due to a consequence of variation in study methodologies, the crude prevalence rate above 60 year-old is 1%. Increase in aging population will lead to an increase in PD patients. The PDR will be used to facilitate the understanding of basic epidemiological features of the disease, genetic and non-genetic risk factors, co-morbidity, the up-to-date treatment strategies and the related economic burden from medical and surgical treatment (deep brain stimulation), to develop new therapeutic protocols as well as healthcare policies, and ultimately, to improve the quality of life of PD patients. PDR will also be served as data bank for investigators in the field of PD to quickly identify and notify research subjects about other research studies for which they are eligible. Patient who registered can also sign their consent for a future brain donation after they passed away.

Methods:

The 4 main Tzu Chi Hospitals from Hualien, Da Lin, Taichung, and Taipei will serve as representative of pilot study for National registry. This will be a record-based, multi-center, nation-wide, cohort study. A user-friendly, yet, encrypted registration platform will be provided through internet for authorized personnel. The contents of PDR will be as follow: demographic features, risk factors, clinical profiles of diagnostic criteria, co-morbidity, images profiles, treatment regimens in details, prognosis, health-related quality of life, and neuropsychological assessment batteries.

Expected results:

1. To facilitate the understanding of demographic epidemiological features of PD.
2. To find the risk factors of PD and the possible intervention toward disease prevention in Taiwan.
3. To find the comorbidity of the disease, and the solution toward better treatment and related outcome.
4. Assess current treatment approaches and develop best-practice guidelines.
5. Tracking the health-related quality of life of PD patient as well as care-givers and the economic impact from different treatment regimens of best medications versus surgical interventions (neuromodulation / neuro-regeneration) from time to time.
6. Drive the development of innovative research projects.
7. Accelerate the process of informing patients of research projects for which they may be eligible.

Key words: Parkinson's disease, Registry, Epidemiology, Treatment, Prognosis

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease

Exclusion Criteria:

* None

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in community hospitals or medical centers
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Risk factors | 1 year
  risk factors include: pesticide, herbicide, drinking underground water, jobs with heavy metals exposure, tea drinking, coffee drinking, smoking, vegetarian

SECONDARY OUTCOMES:
Motor function | 1 year
  Assessment with Unified Parkinson's Disease Rating Scale (UPDRS) part 3. Rating when l-dopa medication On and Off, to see the improvement %.

OTHER OUTCOMES:
Cognitive function | 1 year
  Rating with Mini-mental status examination (MMSE) and Cognitive abilities screening instrument (CASI)
Quality of life | 1 year
  Assessment with Parkinson disease questionnaire (PDQ-39), UPDRS part 2, and Schwab and England activity of daily living (SEADL)
Depression | 1 year
  Assessment with Beck's depression inventory (BDI) and UPDRS part 1.
Comorbidity | 1 year
  Hypertension, diabetes mellitus, stroke, cardiovascular disease, alcoholism, epilepsy, brain surgery, memory impairment, hallucination.
Cost of medical treatment | 1 year
  Identify individual medications and represented as levo-dopar equivalent daily dose (LEDD)
Initial PD symptoms | 1 year
  To identify the initial cardinal symptom: bradykinesia, tremor, rigidity and posture instability

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Yuan Chen, M.D., Principal Investigator — Department of Neurosurgery, Hualien Tzu Chi Hospital
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan